CLINICAL TRIAL: NCT03863392
Title: Oral Misoprostol Solution in Comparison to Vaginal Misoprostol in Induction of Labor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Peter rafik helmy thabet, Clinical investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: test123
Record Dates: First submitted 2019-02-18; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Normal Vaginal Delivery
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- oral (Experimental): patients undergoing induction of labour using misoprostol oral solution
  Interventions: Drug: Misoprostol
- vaginal (Experimental): patients undergoing induction of labour using vaginal misoprostol
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — induction of labor

SUMMARY:
Induction of labour at term is a common obstetric intervention. Induction of labour is the artificial initiation of labour before its spontaneous onset for the purpose of delivery of the fetoplacental unit using mechanical or pharmacological methods.

To determine the effects of oral misoprostol solution compared to vaginal misoprostol in induction of labour.

DETAILED DESCRIPTION:
Patients recruited in the study will be primigravida at term with obstetric or medical indication for labour induction. These patients will be either booked attending antenatal clinic referred for induction of labour or emergency admissions in labour room.

A total of 100 women will be randomly selected for the study. I. Women will be given 20 ml (20 µg) of misoprostol solution orally every 2 hourly until adequate uterine contractions occurred (3 contractions per 10 min lasting 30-40 s).

II. The induction regimen included application of Vagiprost 25 µg tablet in the posterior fornix of the vagina every 4 h (up to 6 doses) after determination of the Bishop score.

ELIGIBILITY:
Inclusion Criteria:

* Primigravida or Primipara
* Pregnancy between 36 and 42 weeks of gestation.
* A live singleton fetus in cephalic presentation.
* No history of uterine surgery.
* Clinically adequate pelvis.
* Modified Bishop's score <5.
* Reactive Non stress test (NST) .

Exclusion Criteria:

* •Known hypersensitivity or contraindications to oral misoprostol (uterine surgery).

  * Any antenatal medical complications.
  * A situation requiring LSCS (Maternal or Fetal) e.g:fetal distress
  * Non-reactive NST.
  * Patient's refusal to give consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2019-03-15 (Estimated)

PRIMARY OUTCOMES:
•Induction-delivery time | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided